CLINICAL TRIAL: NCT00654979
Title: A Pivotal Study to Evaluate the Safety and Effectiveness of RMT Medical Technology's SafeFlo® Vena Cava Filter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RMT Medical Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SFF-104
Record Dates: First submitted 2008-03-30; First posted 2008-04-09 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): SafeFlo IVC Filter
  Interventions: Device: SafeFlo IVC Filter

INTERVENTIONS:
Device: SafeFlo IVC Filter — SafeFlo IVC Filter

SUMMARY:
To determine the safety and effectiveness of the SafeFlo filter for permanent protection against pulmonary emboli. All patients will be selected to receive the filter according to the stated inclusion / exclusion criteria after consultation between the attending physician and interventional radiologist. Patients with a permanent implantation will be followed for up to 6 months. Clinical success will be defined as no occurrences of any of the following events: recurrent pulmonary embolism, IVC occlusion or filter embolization. The proportion of permanent filter patients considered to be a clinical success will be the primary efficacy parameter.

ELIGIBILITY:
Inclusion Criteria:

* Traditional indications for vena cava filter in patients with established DVT or PE, including (40):

  * Patients with proven Pulmonary Embolus (PE) or Deep Vein Thrombosis (DVT) and one or more of the following:

    1. Contraindication to anticoagulation
    2. Complication of anticoagulation
    3. Failure of anticoagulation

       * Recurrent PE despite adequate anticoagulation therapy
       * Inability to achieve adequate anticoagulation
    4. Poor compliance with anticoagulation medications
* Extended indications for vena cava filter placement in patients with established DVT or PE, including the following (31, 40):

  * Large free-floating thrombus in the iliac vein or IVC;
  * Following massive PE in which recurrent emboli may prove fatal;
  * During/after surgical or transcatheter embolectomy;
  * Filter placement in high-risk trauma and orthopedic patients:
* High risk trauma or orthopedic patients who cannot receive anticoagulation because of increased bleeding risk, and have one or more of the following injury patterns (31, 40):

  1. Severe closed head injury (GCS < 8);
  2. Incomplete spinal cord injury with para or quadriplegia;
  3. Complex pelvic fractures with associated long-bone fractures;
  4. Multiple long bone fractures.
* Patients undergoing long-term immobilization (e.g., ICU or Surgical oncology)

Exclusion Criteria:

* All patients under 18 years of age.
* All patients undergoing emergency procedures.
* All patients with abnormal IVC anatomy or pathology of the IVC such as thrombosis or tumor which prevent safe filter implantation.
* All patients with an IVC diameter which precludes oversizing of the filter platform.
* All patients with active infection / bacteremia.
* All patients with sensitivity to contrast media.
* Uncorrectable severe coagulopathy (e.g., patients with liver or multisystem failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2003-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Clinical success will be defined as no occurrences of any of the following events: recurrent pulmonary embolism, IVC occlusion or filter embolization. | 6 months follow-up

SECONDARY OUTCOMES:
The proportion of patients with successful deployment of the filter will be calculated and presented with a 95% exact confidence interval. | 3 and 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Cynamon, Dr., Principal Investigator — Montefiore Medical Center
Locations (8):
- United States (3):
  - Holy Name Hospital, Teaneck, New Jersey
  - Mt. Sinai Hospital, Manhattan, New York
  - Montefiore Medical Center, The Bronx, New York
- University Hospital Vienna, Vienna, Austria
- 251 Air Force Hospital, Athens, Greece
- Rabin Medical Center, Petah Tikva, Israel
- Universitas Hospital, Bloemfontein, South Africa
- Queen Margaret Hospital, Dumfermline, Scotland, United Kingdom

REFERENCES:
- See also: Sponsor Website — http://www.rafaelmedical.com